CLINICAL TRIAL: NCT01360827
Title: Phase Ib Trial of Multiple-ascending Doses of EMD 1201081 in Combination With 5-FU/Cisplatin and Cetuximab in First-line Subjects With Recurrent/ Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: EMD 1201081 + 5-FU + Cisplatin + Cetuximab in Subjects With Recurrent / Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to potential safety concerns in combination with platinum-based therapies
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200068-007
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Safety; tolerability; maximum tolerated dose of EMD 1201081; TLR9 agonists; squamous cell carcinoma of the head and neck; First line subjects; recurrent/metastatic
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis | interventions — IMO-2055; Fluorouracil; Cisplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Part 1) (Experimental)
  Interventions: Drug: EMD 1201081 + 5-FU + Cisplatin + Cetuximab
- Arm 2 (Expansion cohorts -Part 2 and Part 2a) (Experimental)
  Interventions: Drug: EMD 1201081 + 5-FU + Cisplatin + Cetuximab

INTERVENTIONS:
Drug: EMD 1201081 + 5-FU + Cisplatin + Cetuximab — 3-6 subjects per cohort will receive EMD 1201081 as a weekly subcutaneous injection on Days 1, 8, and 15 in 3-week cycles at dose levels of 0.16, 0.32, and 0.48mg/kg, respectively until progression of disease, unacceptable toxicity, or subject refusal to continue in the trial. EMD 1201081 will always be given after (within 1 hour) completion of the cetuximab infusion and before the start of chemotherapy.
  Arms: Arm 1 (Part 1)
Drug: EMD 1201081 + 5-FU + Cisplatin + Cetuximab — Part 2 seeks to enroll 12 subjects at the MTD of EMD 1201081 in combination with 5-FU/cisplatin + cetuximab; furthermore, an additional 3 to 6 subjects for a total of 9 subjects will be accrued at the 0.16 mg/kg low dose level in Part 2a once the Part 1 0.16 mg/kg dose cohort has been accrued and it is deemed safe to proceed to the 0.32 mg/kg dose cohort. EMD 1201081 will always be given after (within 1 hour) completion of the cetuximab infusion and before the start of chemotherapy.
  Arms: Arm 2 (Expansion cohorts -Part 2 and Part 2a)

SUMMARY:
The primary purpose of this trial is to assess the safety and tolerability of EMD 1201081, a novel immunomodulatory agent that is an agonist of TLR9, in combination with 5-FU/cisplatin and cetuximab in first line treatment of patients with recurrent/metastatic squamous cell carcinoma of the head and neck, and to determine the maximum tolerated dose (MTD) among the dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of squamous cell carcinoma of the head and neck (SCCHN).
* Recurrent and/or metastatic SCCHN, not suitable for local therapy.
* At least 1 measurable lesion either by computerized tomography (CT) scan or magnetic resonance imaging (MRI) (according to RECIST 1.0).
* Karnofsky performance status (KPS) of ≥ 70 / Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1 at trial entry.

Exclusion Criteria:

* Prior systemic chemotherapy, except if given as part of a multimodal treatment for locally advanced disease which was completed more than 2 months prior to trial entry.
* Nasopharyngeal carcinoma.
* Medical history of diagnosed interstitial lung disease.
* Known hypersensitivity against any of the components of the trial treatment.
* Previous treatment with experimental or non-approved epidermal growth factor receptor (EGFR) targeting therapy or experimental or nonapproved EGFR signal transduction inhibitors (prior treatment with cetuximab is allowed).
* Relevant cardiovascular co-morbidities.
* Concomitant chronic systemic immune therapy, or hormonal therapy as cancer therapy, steroid use ≥ 10 mg prednisone equivalent.
* Known human immunodeficiency virus (HIV) positivity, active hepatitis C, or active hepatitis B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated-dose (MTD) at 0.16 mg/kg cohort size testing | 3 weeks
  Occurrence of treatment-related dose-limiting toxicity during the first cycle (3 weeks) of treatment in subjects treated with multi-ascending doses of EMD 1201081 in combination with 5-FU/cisplatin + cetuximab.
Maximum-tolerated-dose (MTD) at 0.32 mg/kg cohort size testing | 3 weeks
  Occurrence of treatment-related dose-limiting toxicity during the first cycle (3 weeks) of treatment in subjects treated with multi-ascending doses of EMD 1201081 in combination with 5-FU/cisplatin + cetuximab.
Maximum-tolerated-dose (MTD) at 0.48 mg/kg cohort size testing | 3 weeks
  Occurrence of treatment-related dose-limiting toxicity during the first cycle (3 weeks) of treatment in subjects treated with multi-ascending doses of EMD 1201081 in combination with 5-FU/cisplatin + cetuximab.
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | Baseline up to 49 days after last study drug administration

SECONDARY OUTCOMES:
Number of subjects with best overall response | 8 months
Pharmacokinetic parameters: Cmax, Tmax and AUC (0-t) | Days 1, 8 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jean-Pierre Delord, Principal Investigator — Clinical Research Unit and Pharmacology Lab EA 3035, Institut Claudius Regaud, Toulouse, France
Locations (1):
- Clinical Research Unit and Pharmacology Lab EA 3035 Institut Claudius Regaud, Toulouse, France